CLINICAL TRIAL: NCT01674712
Title: A 12-week, Double-blind, Randomized Study to Compare the Efficacy and Safety of Fixed Combinations of Fenofibrate / Simvastatin 145/20mg and Fenofibrate / Simvastatin 145/40mg Tablets vs. Matching Monotherapies in Dyslipidemic Subjects at High Risk of Cardiovascular Disease.
Brief Title: A 12-week Study to Compare the Efficacy and Safety of Fixed Combinations of Fenofibrate/Simvastatin 145/20mg and Fenofibrate/Simvastatin 145/40mg Tablets Versus Fenofibrate or Simvastatin Monotherapies in Subjects With Abnormal Blood Levels of Fats (Lipids) and at High Risk of Cardiovascular Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Abbott (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: M13-377; 2011-005924-16 (EudraCT Number)
Record Dates: First submitted 2012-06-26; First posted 2012-08-29 (Estimated); Results first posted 2014-10-30 (Estimated); Last update posted 2014-12-11 (Estimated); Status verified 2014-11

CONDITIONS: Dyslipidemia
Keywords: Fibrates; Dyslipidemia
MeSH Terms: conditions — Dyslipidemias | interventions — Simvastatin; Fenofibrate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor

ARMS (5):
- Fenofibrate/simvastatin 145/20 mg (Experimental)
  Interventions: Drug: Fixed Combination of Fenofibrate/simvastatin 145/20 mg
- Simvastatin 20 mg (Active Comparator)
  Interventions: Drug: Simvastatin 20 mg
- Fenofibrate 145 mg (Active Comparator)
  Interventions: Drug: Fenofibrate 145 mg
- Fenofibrate/simvastatin 145/40 mg (Experimental)
  Interventions: Drug: Fixed Combination of Fenofibrate/simvastatin 145/40 mg
- Simvastatin 40 mg (Active Comparator)
  Interventions: Drug: Simvastatin 40 mg

INTERVENTIONS:
Drug: Fixed Combination of Fenofibrate/simvastatin 145/20 mg — Fenofibrate/simvastatin oval biconvex film-coated tablet, 145 mg / 20 mg, once daily, 12 weeks
  Arms: Fenofibrate/simvastatin 145/20 mg
Drug: Simvastatin 20 mg — Simvastatin generic tablet over-encapsulated, 20 mg, once daily, 12 weeks
  Arms: Simvastatin 20 mg
Drug: Fenofibrate 145 mg — Fenofibrate, tablet, 145 mg, once daily, 12 weeks
  Arms: Fenofibrate 145 mg
Drug: Fixed Combination of Fenofibrate/simvastatin 145/40 mg — Fenofibrate/simvastatin film-coated tablet 145 mg / 40 mg, once daily, 12 weeks
  Arms: Fenofibrate/simvastatin 145/40 mg
Drug: Simvastatin 40 mg — simvastatin, generic tablet over-encapsulated, 40 mg, once daily, 12 weeks
  Arms: Simvastatin 40 mg

SUMMARY:
This is a double-blind, randomized study designed to compare the efficacy and safety of two fixed combinations of fenofibrate / simvastatin 145/20 mg and fenofibrate / simvastatin 145/40 mg tablets vs. matching monotherapies in subjects with abnormal fat (lipids) in the blood and at high risk of cardiovascular disease. Fenofibrate is a treatment that lowers fat in blood. It is prescribed in patients with high levels of triglycerides (TG). The drug has been marketed in more than 80 countries since 1975. Simvastatin is also used for the treatment of patients with a high level of cholesterol. These have also been marketed worldwide for more than 20 years. It is important to treat high levels of fats in the blood because it has been shown that even mildly elevated level of lipids in the blood can lead to diseases of the blood vessels. It has been shown in several studies and in clinical practice that the combination of fenofibrate plus simvastatin can lead to improved effects on blood fats, compared to treatment with simvastatin or fenofibrate alone. The main objective of the study is to compare the efficacy of the two fixed-combinations (FC) -fenofibrate/simvastatin 145/20 mg tablet and fenofibrate/simvastatin 145/40 mg tablet in reducing TG and increasing high density lipoprotein cholesterol (HDL-C) versus simvastatin 20 mg or 40 mg, and in reducing low density lipoprotein cholesterol (LDL-C) versus fenofibrate 145 mg.

ELIGIBILITY:
Inclusion Criteria:

1. Either gender (tentatively 50 percent females to be included and if of childbearing potential she must agree to use medically acceptable methods of contraception from the time of signing the informed consent until 7 days following administration of the last treatment or dose of study medication). Accepted contraceptive methods are implants, injectables, combined oral contraceptives, intra-uterine device or sexual abstinence.
2. between 18 (inclusive) and 80 years
3. With mixed dyslipidemia with fasting lipid results of a blood sample taken at inclusion and after at least 3 months of any statin monotherapy (excluding simvastatin 80 mg, atorvastatin 40 mg and 80 mg, rosuvastatin 20 mg and 40 mg):

   * TG higher than/equal to 1.71 mmol/L (higher than/equal to 150 mg/dL) and
   * LDL-C higher or equal to 1.81 mmol/L (higher or equal 70 mg/dL) but smaller than/equal to 3.36 mmol/L (smaller than/equal to 130 mg/dL)
4. High risk or very high risk based on known CardioVascular Disease (CVD) or type 2 diabetes or type 1 diabetes with microalbuminuria or a Systematic Coronary Risk Estimation (SCORE) chart risk ≥ 5percent
5. Aspartate aminotransferase and/or alanine aminotransferase smaller than/equal to 2 times the Upper Normal of Limit (UNL)

Exclusion Criteria:

1. Known hypersensitivity to fibrates or simvastatin or known photoallergic or phototoxic reactions under treatment with fibrates or ketoprofen or known allergic reactions caused by peanuts, peanuts or arachis oil or soy lecithin, or related products,
2. Pregnant or lactating women,
3. Unable or unwilling to comply with the protocol and the recommended diet,
4. Likely to withdraw from the study before its completion,
5. Having received an investigational drug or vaccine in the last 30 days before date of inclusion, or still participating in such a trial at Visit 1

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 575 (Actual)
Dates: Start 2012-06; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jean-Claude Ansquer, MD, Study Director — Abbott
Locations (69):
- Argentina (15):
  - Site Reference ID/Investigator# 77961, Buenos Aires
  - Site Reference ID/Investigator# 77957, Buenos Aires
  - Site Reference ID/Investigator# 77958, Buenos Aires
  - Site Reference ID/Investigator# 77960, Buenos Aires
  - Site Reference ID/Investigator# 77959, Buenos Aires
  - Site Reference ID/Investigator# 77969, Buenos Aires
  - Site Reference ID/Investigator# 77967, Buenos Aires
  - Site Reference ID/Investigator# 77968, Buenos Aires
  - Site Reference ID/Investigator# 77965, Buenos Aires
  - Site Reference ID/Investigator# 77956, Buenos Aires
  - Site Reference ID/Investigator# 77966, Cipolletti - Rio Negro
  - Site Reference ID/Investigator# 77963, San Miguel de Tucumán
  - Site Reference ID/Investigator# 77955, Santa Fe
  - Site Reference ID/Investigator# 77962, Santa Fe
  - Site Reference ID/Investigator# 77964, Santa Fe
- Czechia (9):
  - Site reference ID/Investigator # 99617, Benátky nad Jizerou
  - Site Reference ID/Investigator# 80097, Brno
  - Site reference ID/Investigator # 102335, Brno
  - Site Reference ID/Investigator# 80094, Prague
  - Site Reference ID/Investigator# 80095, Prague
  - Site Reference ID/Investigator# 80093, Prague
  - Site Reference ID/Investigator# 80098, Teplice
  - Site Reference ID/Investigator# 80096, Ústí nad Labem
  - Site Reference ID/Investigator# 80099, Znojmo
- Germany (14):
  - Site reference ID/Investigator # 97356, Berlin
  - Site Reference ID/Investigator# 90673, Berlin
  - Site Reference ID/Investigator# 80100, Berlin
  - Site reference ID/Investigator # 97357, Berlin
  - Site reference ID/Investigator # 102016, Cologne
  - Site reference ID/Investigator # 102017, Dortmund
  - Site reference ID/Investigator # 99876, Dresden
  - Site Reference ID/Investigator# 80102, Düsseldorf
  - Site Reference ID/Investigator# 80104, Essen
  - Site Reference ID/Investigator# 80103, Essen
  - Site Reference ID/Investigator# 80105, Frankfurt
  - Site Reference ID/Investigator# 80101, Goch
  - Site reference ID/Investigator # 99902, Hamburg
  - Site reference ID/Investigator # 102015, Karlsruhe
- Mexico (4):
  - Site Reference ID/Investigator# 77970, Guadalajara, Jal.
  - Site Reference ID/Investigator# 77973, Mexico City
  - Site Reference ID/Investigator# 77972, Mexico City
  - Site Reference ID/Investigator# 77974, Zapopan
- Poland (7):
  - Site Reference ID/Investigator# 80111, Gdansk
  - Site Reference ID/Investigator# 80112, Gdansk
  - Site Reference ID/Investigator# 80110, Gdynia
  - Site Reference ID/Investigator# 80106, Katowice
  - Site Reference ID/Investigator# 80109, Płock
  - Site Reference ID/Investigator# 80108, Skierniewice
  - Site Reference ID/Investigator# 80107, Warsaw
- Romania (7):
  - Site reference ID/Investigator # 80115, Bucharest
  - Site Reference ID/Investigator# 80114, Bucharest
  - Site Reference ID/Investigator# 80117, Bucharest
  - Site Reference ID/Investigator# 80116, Bucharest
  - Site Reference ID/Investigator# 80119, Bucharest
  - Site Reference ID/Investigator# 80113, Bucharest
  - Site Reference ID/Investigator# 80118, Iași
- Russia (13):
  - Site Reference ID/Investigator# 80120, Kemerovo
  - Site Reference ID/Investigator# 80135, Moscow
  - Site Reference ID/Investigator# 80137, Moscow
  - Site Reference ID/Investigator# 80124, Moscow
  - Site Reference ID/Investigator# 80127, Moscow
  - Site Reference ID/Investigator# 80122, Novosibirsk
  - Site Reference ID/Investigator# 80121, Novosibirsk
  - Site Reference ID/Investigator# 80133, Novosibirsk
  - Site reference ID/Investigator # 80134, Saint Petersburg
  - Site reference ID/Investigator # 80126, Saint Petersburg
  - Site reference ID/Investigator # 80128, Saint Petersburg
  - Site Reference ID/Investigator# 80136, Saint Petersburg
  - Site Reference ID/Investigator# 80125, Yaroslavl

RESULTS

PARTICIPANT FLOW:
Groups:
- Fenofibrate/Simvastatin 145/20 mg: Fenofibrate/simvastatin 145/20 mg: Fenofibrate/simvastatin oval biconvex film-coated tablet, 145 mg / 20 mg, once daily, 12 weeks
- Fenofibrate/Simvastatin 145/40 mg: Fenofibrate/simvastatin 145/40 mg: Fenofibrate/simvastatin film-coated tablet 145 mg / 40 mg, once daily, 12 weeks
Period: Overall Study
Arm/Group | Fenofibrate/Simvastatin 145/20 mg | Simvastatin 20 mg | Fenofibrate/Simvastatin 145/40 mg | Simvastatin 40 mg | Fenofibrate 145 mg
Started | 114 | 117 | 115 | 116 | 113
Full Analysis Subject Sample | 109 | 114 | 110 | 112 | 111
Safety Subject Sample | 111 | 117 | 113 | 115 | 112
Completed | 104 | 108 | 106 | 108 | 102
Not Completed | 10 | 9 | 9 | 8 | 11
Not completed — Adverse Event | 5 | 6 | 3 | 4 | 6
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0 | 0
Not completed — Protocol Violation | 2 | 0 | 0 | 0 | 0
Not completed — Withdrawal by Subject | 2 | 2 | 5 | 4 | 3
Not completed — Administrative | 0 | 1 | 0 | 0 | 1
Not completed — Lack of Efficacy | 0 | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Full analysis subject sample
Groups:
- Total: Total of all reporting groups
Arm/Group | Fenofibrate/Simvastatin 145/20 mg | Simvastatin 20 mg | Fenofibrate/Simvastatin 145/40 mg | Simvastatin 40 mg | Fenofibrate 145 mg | Total
Number analyzed (Participants) | 109 | 114 | 110 | 112 | 111 | 556
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.6 (10) | 60.5 (9.3) | 60.4 (8.1) | 59.3 (9.1) | 60.4 (9.0) | 60.0 (9.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 38 | 40 | 43 | 39 | 38 | 198
  Male | 71 | 74 | 67 | 73 | 73 | 358
Region of Enrollment [Number; unit: participants]
  Czech Republic | 22 | 22 | 22 | 23 | 21 | 110
  Mexico | 7 | 9 | 8 | 7 | 8 | 39
  Argentina | 19 | 22 | 19 | 20 | 21 | 101
  Poland | 7 | 9 | 8 | 10 | 7 | 41
  Romania | 6 | 6 | 6 | 5 | 4 | 27
  Russian Federation | 18 | 17 | 16 | 16 | 17 | 84
  Germany | 30 | 29 | 31 | 31 | 33 | 154
Triglycerides (mmol/L) [Mean (Standard Deviation); unit: mmol/L] | 2.8 (1.1) | 2.5 (1.0) | 2.7 (1.4) | 2.7 (1.0) | 2.9 (1.3) | 2.7 (1.1)
LDL Cholesterol (mmol/L) [Mean (Standard Deviation); unit: mmol/L] | 2.6 (0.5) | 2.6 (0.4) | 2.6 (0.4) | 2.7 (0.4) | 2.7 (0.5) | 2.7 (0.5)
HDL Cholesterol (mmol/L) [Mean (Standard Deviation); unit: mmol/L] | 1.1 (0.3) | 1.2 (0.3) | 1.2 (0.3) | 1.2 (0.3) | 1.2 (0.3) | 1.2 (0.3)

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Change of TG (Triglyceride)
Description: Collection and measurement of blood samples.
Time Frame: from baseline to 12 weeks of treatment
Population: The Primary Analysis was done for the sample set of patients with 12 weeks' assessment.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Fenofibrate/Simvastatin 145/20 mg | Simvastatin 20 mg | Fenofibrate/Simvastatin 145/40 mg | Simvastatin 40 mg | Fenofibrate 145 mg
Number analyzed (Participants) | 96 | 102 | 97 | 101 | 93
percentage of change | -30.6 (25.8) | 10.7 (48.8) | -27.3 (35.9) | -2.9 (34.3) | -21.6 (34.2)

2. Primary Outcome: Percentage of Change of HDL-C (High Density Lipoprotein Cholesterol)
Description: Collection and measurement of blood samples.
Time Frame: from baseline to 12 weeks of treatment
Population: The Primary Analysis was done for the sample set of patients with 12 weeks' assessment.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Fenofibrate/Simvastatin 145/20 mg | Simvastatin 20 mg | Fenofibrate/Simvastatin 145/40 mg | Simvastatin 40 mg | Fenofibrate 145 mg
Number analyzed (Participants) | 96 | 102 | 97 | 101 | 93
percentage of change | 9.0 (16.8) | 0.3 (12.1) | 8.8 (16.5) | 2.2 (12.5) | 7.6 (15.7)

3. Primary Outcome: Percentage of Change of LDL-C (Low Density Lipoprotein Cholesterol)
Description: Collection and measurement of blood samples.
Time Frame: from baseline to 12 weeks of treatment
Population: The Primary Analysis was done for the sample set of patients with 12 weeks' assessment.
Measure: Mean (Standard Deviation); unit: percentage of change
Arm/Group | Fenofibrate/Simvastatin 145/20 mg | Simvastatin 20 mg | Fenofibrate/Simvastatin 145/40 mg | Simvastatin 40 mg | Fenofibrate 145 mg
Number analyzed (Participants) | 96 | 102 | 97 | 101 | 93
percentage of change | 1.9 (25.4) | -2.0 (24.8) | -6.1 (26.2) | -8.1 (25.8) | 30.3 (35.6)

4. Secondary Outcome: Percentage of Non-HDL (High Density Lipoprotein)-C From Baseline
Description: Collection and measurement of blood samples
Time Frame: 12 weeks
Reporting Status: Not Posted

5. Secondary Outcome: Percentage of TC (Triglyceride) From Baseline
Description: Collection and measurement of blood samples
Time Frame: 12 weeks
Reporting Status: Not Posted

6. Secondary Outcome: Percentage of Apolipoprotein AI From Baseline
Description: Collection and measurement of blood samples
Time Frame: 12 weeks
Reporting Status: Not Posted

7. Secondary Outcome: Percentage of Apolipoprotein B From Baseline
Description: Collection and measurement of blood samples
Time Frame: 12 weeks
Reporting Status: Not Posted

8. Secondary Outcome: Percentage of High-sensitivity C-reactive Protein (hsCRP) From Baseline
Description: Collection and measurement of blood samples
Time Frame: 12 weeks
Reporting Status: Not Posted

9. Secondary Outcome: Percentage of Subjects Meeting Target Levels of Lipids (According to Very High or High Risk)
Description: Collection and measurement of blood samples
Time Frame: 12 weeks
Reporting Status: Not Posted

10. Secondary Outcome: Adverse Events
Description: Collection and measurement of blood samples
Time Frame: 12 weeks
Reporting Status: Not Posted

11. Secondary Outcome: Creatine Kinase (CK)
Description: Collection and measurement of blood samples
Time Frame: 12 weeks
Reporting Status: Not Posted

12. Secondary Outcome: Alanine Aminotransferase (ALT)
Description: Collection and measurement of blood samples
Time Frame: 12 weeks
Reporting Status: Not Posted

13. Secondary Outcome: Plasma Creatinine
Description: Collection and measurement of blood samples
Time Frame: 12 weeks
Reporting Status: Not Posted

14. Secondary Outcome: Total Bilirubin
Description: Collection and measurement of blood samples
Time Frame: 12 weeks
Reporting Status: Not Posted

15. Secondary Outcome: Cystatin C
Description: Collection and measurement of blood samples
Time Frame: 12 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Arm/Group | Fenofibrate/Simvastatin 145/20 mg | Simvastatin 20 mg | Fenofibrate/Simvastatin 145/40 mg | Simvastatin 40 mg | Fenofibrate 145 mg
Serious Adverse Events (participants affected / at risk) | 3/111 | 3/117 | 3/113 | 1/115 | 3/112
Other Adverse Events (participants affected / at risk) | 8/111 | 7/117 | 4/113 | 9/115 | 15/112
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Fenofibrate/Simvastatin 145/20 mg (N=111) | Simvastatin 20 mg (N=117) | Fenofibrate/Simvastatin 145/40 mg (N=113) | Simvastatin 40 mg (N=115) | Fenofibrate 145 mg (N=112)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
ACUTE MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
ANGINA PECTORIS (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) — One Myocardial Infarction was fatal.
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
DIABETES MELLITUS INADEQUATE CONTROL (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
CEREBROVASCULAR ACCIDENT (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
LOSS OF CONSCIOUSNESS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
INTESTINAL HAEMORRHAGE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
UMBILICAL HERNIA, OBSTRUCTIVE (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
NON-SITE SPECIFIC INJURIES NEC (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) — One Injury was fatal.
BURSITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
HAEMATURIA (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
DIABETES MELLITUS MANAGEMENT (Surgical and medical procedures) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Fenofibrate/Simvastatin 145/20 mg (N=111) | Simvastatin 20 mg (N=117) | Fenofibrate/Simvastatin 145/40 mg (N=113) | Simvastatin 40 mg (N=115) | Fenofibrate 145 mg (N=112)
DIARRHOEA (Gastrointestinal disorders) | 1 | 2 | 2 | 0 | 5
NASOPHARYNGITIS (Infections and infestations) | 1 | 0 | 1 | 3 | 3
BLOOD CREATINE PHOSPHOKINASE INCREASED (Investigations) | 4 | 0 | 1 | 1 | 1
GASTROENTERITIS (Infections and infestations) | 1 | 2 | 0 | 0 | 4
DYSPEPSIA (Gastrointestinal disorders) | 1 | 0 | 0 | 4 | 1
COUGH (Respiratory, thoracic and mediastinal disorders) | 0 | 3 | 0 | 1 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
At least sixty (60) days prior to submitting or presenting a manuscript or other materials relating to the Study to a publisher, reviewer, or other outside persons, the PI shall provide to Sponsor a copy of all such manuscripts and materials, and allow Sponsor sixty (60) days to review and comment on them. If the Sponsor requests, the PI shall remove any Confidential Information (other than Study results) prior to submitting or presenting the materials.